CLINICAL TRIAL: NCT02771899
Title: Value of 3D Modeling in Spine Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor and PI decision
Sponsor: Columbia University (Other)
Collaborators: EOS imaging Inc. (Industry)
Responsible Party: Principal Investigator, Lawrence Lenke, Professor of Orthopedic Surgery at the Columbia University Medical Center, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAQ6551
Record Dates: First submitted 2016-05-07; First posted 2016-05-13 (Estimated); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Scoliosis
Keywords: Imaging, Three-Dimensional; Spine; Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- EOS + spineEOS software in adults (Experimental): Participants will receive standard of care (EOS) - 2D planning with 3D modeling.
  Interventions: Device: spineEOS software; Device: EOS
- EOS in adults (Active Comparator): Participants will receive standard of care (EOS) - 2D planning performed with current practice.
  Interventions: Device: EOS
- EOS + spineEOS software in children (Experimental): Participants will receive standard of care (EOS) - 2D planning with 3D modeling.
  Interventions: Device: spineEOS software; Device: EOS
- EOS in children (Active Comparator): Participants will receive standard of care (EOS) - 2D planning performed with current practice.
  Interventions: Device: EOS

INTERVENTIONS:
Device: spineEOS software — During a full-length exam from head to feet in the standing position, 3D reconstructions of the spine, the pelvis and lower extremities using spine workflow and global postural assessment workflow on spineEOS software will be performed.
  Other Names: 3D spine reconstructions; 3D Modeling; spineEOS workstation
  Arms: EOS + spineEOS software in adults; EOS + spineEOS software in children
Device: EOS — The system performs a full-length exam from head to feet in the standing position. 2D parameters will be obtained per standard of care.
  Other Names: biplanar low-dose EOS system; 2D Planning

SUMMARY:
Adults (18 years and over) and children (10-17 years of age) scheduled for surgery to correct scoliosis will be included in this study, for which participation will last 6 months. Each age group of participants will be randomized to two cohorts: one cohort will receive standard of care, while the other will also have their standard radiographic images used in the construction of a three-dimensional visualization of the spine. Questionnaires administered before and after surgery, in addition to health information collected throughout the course of the study, will indicate whether the three-dimensional model has an effect on the planning, performance, and outcomes of surgery. Participants in this study will not be asked to do anything outside the standard of care. The only manipulated variable in this study is the construction of the three dimensional model, which is made from information collected during the standard of care, and requires no further action on the participant's behalf. The results of this study may show that three-dimensional visualizations can be of value to spinal surgeons, and positively affect patient outcomes.

DETAILED DESCRIPTION:
The biplanar low-dose EOS system and its associated spineEOS workstation (EOS®, EOS Imaging, Paris, France) allows 3D spine reconstructions. The EOS system presents some advantages over MRI or CT Scans. The weight bearing position allows assessment in the functional position and the radiation exposure is 800-1000 times less then CT scans, allowing full spine acquisition even in pediatric patients. Selected anatomical landmarks are utilized to reconstruct a 3D model of the spine allowing global assessment as well as localized analysis.The aim of the study is to assess the clinical relevance of 3D stereographic reconstructions (from spineEOS 3D) on patients, adults and children, who undergo spine surgery. This study will observe the value of 3D parameters at three different steps of the standard of care surgical procedure: preoperatively, peri-operatively, and post-operatively. The goal of this prospective study is to observe how 3D reconstructions could enhance the planning, the surgery and the post-op analysis and outcomes. This pilot study could help to understand which and how 3D parameters could improve adult and pediatric spine surgery.

ELIGIBILITY:
Adults --

Inclusion Criteria:

* All patients must be age 18 or greater at the time of surgery or initial consultation
* Having a primary surgery of their spine (fusion or instrumentation)

Exclusion Criteria:

* Diagnosis of scoliosis other than degenerative or idiopathic (i.e., paralytic/neuromuscular, congenital)
* Undergoing revision (fusion or instrumentation)

EOS Exclusion Criteria:

* Patients with supernumerary vertebrae (one extra or one less thoracic or lumbar vertebrae)
* Insufficient quality of images to perform the 3D modeling with spineEOS software

Children --

Inclusion Criteria:

* All patients must be younger than 18 at the time of surgery
* Having a primary surgery of their spine (fusion or instrumentation)

Exclusion Criteria:

* Diagnosis of scoliosis other than degenerative or idiopathic (i.e., paralytic/neuromuscular, congenital
* Undergoing revision (fusion or instrumentation)

EOS Exclusion Criteria:

* Patients with supernumerary vertebrae (one extra or one less thoracic or lumbar vertebrae)
* Insufficient quality of images to perform the 3D modeling with spineEOS software

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-04-19 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence G Lenke, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EOS + spineEOS Software in Adults | EOS in Adults | EOS + spineEOS Software in Children | EOS in Children
Started | 20 | 17 | 6 | 11
Completed | 0 | 0 | 0 | 0
Not Completed | 20 | 17 | 6 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EOS + spineEOS Software in Adults | EOS in Adults | EOS + spineEOS Software in Children | EOS in Children | Total
Number analyzed (Participants) | 20 | 17 | 6 | 11 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 6 | 11 | 17
  Between 18 and 65 years | 13 | 14 | 0 | 0 | 27
  >=65 years | 7 | 3 | 0 | 0 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (18) | 52 (19.9) | 16 (2.8) | 16 (2) | 38 (21.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 4 | 8 | 34
  Male | 9 | 6 | 2 | 3 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 17 | 6 | 11 | 54

OUTCOME MEASURES:

1. Primary Outcome: Questionnaire Showing the 3D Imaging Helped Surgery Planning
Description: The surgeon will complete a one-question surgical questionnaire regarding their perceptions of the value of 3D modeling brought to the care of their patient. "Did the 3D imaging help with planning the surgery?" Yes = it helped. No = it did not help.
Time Frame: 1 week post-operatively
Population: Only completed questionnaires for 11 subjects were analyzed: 7 out of 20 EOS + spineEOS software in adults and 4 out of 6 EOS + spineEOS software in children had completed questionnaires.
Measure: Count of Participants; unit: Participants
Arm/Group | EOS + spineEOS Software in Adults | EOS + spineEOS Software in Children
Number analyzed (Participants) | 7 | 4
Participants
  Yes | 0 | 0
  No | 7 | 4

2. Secondary Outcome: Health Related Quality Of Life (HRQOL) Score
Description: The standardized Scoliosis Research Society-22r questionnaire consists of 22 questions that assesses the patient's physical function, pain, self-image, mental health, and satisfaction with treatment. The minimum score is 22 and the highest score is 110. A higher score indicates a better outcome.
Time Frame: 3-4 months post-op
Population: Only completed questionnaires for 4 subjects were analyzed: 2 out of 20 EOS + spineEOS software in adults and 2 out of 6 EOS + spineEOS software in children had completed questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EOS + spineEOS Software in Adults | EOS in Adults | EOS + spineEOS Software in Children | EOS in Children
Number analyzed (Participants) | 2 | 0 | 2 | 0
score on a scale | 103 (6) |  | 106 (3) |

ADVERSE EVENTS:
Time Frame: Up to 4 months
Arm/Group | EOS + spineEOS Software in Adults | EOS in Adults | EOS + spineEOS Software in Children | EOS in Children
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/17 | 0/6 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/17 | 0/6 | 0/11
Other Adverse Events (participants affected / at risk) | 0/20 | 0/17 | 0/6 | 0/11

LIMITATIONS AND CAVEATS:
The PI and sponsor decided to end the study early because the spineEOS software did not seem to make a difference in surgery planning.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT02771899/Prot_SAP_000.pdf